CLINICAL TRIAL: NCT03407495
Title: A Phase II, Multi-Center, Open-Label, Single-Arm Study to Evaluate the Clinical Validity and Safety of IOP Injection for Magnetic Resonance Imaging (MRI) Contrast Agent in Hepatocellular Carcinoma (HCC)
Brief Title: The Clinical Validity and Safety of IOP Injection MRI Contrast Agent in Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MegaPro Biomedical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IOP-CT-003
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Magnetic Resonance Imaging
Keywords: Hepatocellular Carcinoma; Magnetic Resonance Imaging
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- single arm: IOP injection (MPB-1523) (Experimental): single group treatment
  Interventions: Drug: IOP Injection (MPB-1523)

INTERVENTIONS:
Drug: IOP Injection (MPB-1523) — one dose, once IV injection at Day 1
  Other Names: MRI Contrast Agent

SUMMARY:
This study is an exploratory study aiming to collect data on sensitivity and positive predictive value of IOP-enhanced (MPB-1523) MRI compared to dynamic multiphase MDCT for the detection of HCC.

DETAILED DESCRIPTION:
The planned duration of the clinical study for individual subjects is up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years of age
2. Patients with suspected HCC scheduled for partial hepatic resection.
3. Presenting with 1 to a maximum of 5 hepatic nodule(s) of equal or more than 1 cm (long axis) previously identified and characterized through multi-phase contrast enhanced CT.
4. Subjects or their partners must use a highly effective method of contraception starting from at least one menstrual cycle prior to starting study drug and till 30 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects who received any previous treatment for HCC.
2. Subjects with a serious allergic history or known allergy of other contrast agent.
3. Subjects with a positive HIV test.
4. Subjects with severe renal insufficiency
5. Subjects with severe liver disease[HCV].
6. Subjects with active systemic infections, active and clinically significant cardiac diseases, active gastrointestinal ulcers, or medical conditions that may significantly affect action, adequate absorption, and elimination of investigational contrast agent.
7. Subject with mechanically, electrically or magnetically-activated implanted device or any metal in their body which cannot be removed.
8. Subjects who have participated in other investigational trials within 30 days prior to study enrollment.
9. Female subjects who are pregnant or breastfeeding.
10. Subjects who are clinically unstable and whose clinical course during the screening period is unpredictable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The Sensitivity and specificity of IOP-enhanced MRI | After IOP injection administration within 60 mins
  Sensitivity and specificity of IOP-enhanced MRI will be calculated using dynamic multiphase MDCT as the reference standard. Confirmation of the diagnosis of HCC lesions will be obtained by surgery.

SECONDARY OUTCOMES:
Optimal time to perform a MRI scan after injection of IOP | After IOP injection administration within 60 mins
  Optimal time of IOP Injection
The Number of lesions detected in liver | After IOP injection administration within 60 mins
  The sensitivity of IOP Injection
The size of lesions detected in liver | After IOP injection administration within 60 mins
  The sensitivity of IOP Injection

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Chen, MD, Principal Investigator — National Taiwan University Hospital; David Wang, MD, Study Director — MegaPro Biomedical Co. Ltd.
Locations (5):
- Taiwan (5):
  - Chang Gung Medical Foundation, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei